CLINICAL TRIAL: NCT06199726
Title: REFLECT: Reproductive Education and Fertility Links for Cancer Treatment
Acronym: REFLECT
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-22569
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Reproductive Behavior
Keywords: Fertility
MeSH Terms: conditions — Reproductive Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Round 1 Interviews and/or Focus Group: Approximately12 people will be recruited complete interviews or focus groups in Round 1.
  The participants will be provided with the REFLECT tool. There will be interviews and discussions via telephone or ZOOM and feedback will be obtained to enhance the REFLECT tool.
  Interventions: Behavioral: REFLECT web-based tool
- Round 2 Interviews and/or Focus Group: Approximately 13 people will be recruited to complete interviews or focus group in Round 2.
  The participants will be provided with the REFLECT tool that has been modified to include feedback from Round 1 interviews/focus groups.
  There will be interviews and discussions via telephone or ZOOM and feedback will be obtained on the enhanced tool.
  Interventions: Behavioral: REFLECT web-based tool

INTERVENTIONS:
Behavioral: REFLECT web-based tool — Partnering with Nest Genomics, Investigators have developed a customizable web-based tool to support AYA patients through their cancer diagnosis journey for topics related to future family building and genetics. This interactive tool will include educational content to organize knowledge, make connections between concepts, and will include web links to more in-depth content and embedded videos. The interface will allow users to document questions that would be helpful in provider discussions and include decision support to assist with determining values and needs for proceeding with consultations related to genetic counseling and testing, and fertility.

SUMMARY:
The purpose of this study is to evaluate a web-based education tool geared at helping Adolescent and Young Adult (AYA) patients better understand fertility and genetic risks for cancer in future offspring.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18-39
* Must have received Cancer care at Moffitt Cancer Center
* Participants must consider having a child in the future or have had children at the time of diagnosis
* Participants must be able to speak and read English
* Participants must have access to a device that can connect to the internet

Exclusion Criteria:

* Any participants who do not meet all Inclusion Criteria

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults ages 18-39 who have received cancer care at Moffitt and have children or are considering having a chilid in the future.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Ease of use of the REFLECT tool | One Year
  System usability scale of 1-5 (1 strongly disagree and 5 strongly agree)
Confidence in use of the REFLECT tool | One Year
  System usability scale of 1-5 (1 strongly disagree and 5 strongly agree)
Complexity of use of the REFLECT tool | One Year
  System usability scale of 1-5 (1 strongly disagree and 5 strongly agree)
Desire to use the REFLECT tool | One Year
  System usability scale of 1-5 (1 strongly disagree and 5 strongly agree)
Perception of inconsistencies of the REFLECT tool | One Year
  System usability scale of 1-5 (1 strongly disagree and 5 strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Vadaparampil, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center's Clinical Trials Website — http://moffitt.org/clinicaltrials